CLINICAL TRIAL: NCT07166185
Title: Evaluation of the Efficacy of Subcutaneous Trastuzumab-Pertuzumab Combination in Neoadjuvant Treatment of Non-Metastatic HER2-Positive Breast Cancer in Algerian Women
Brief Title: Efficacy of Neoadjuvant Subcutaneous Trastuzumab-Pertuzumab in Algerian Women With Locally Advanced HER2 Positive Breast Cancer
Acronym: NEOTRAPSCAL
Status: Recruiting | Type: Observational
Sponsor: Blida 1 University (Other)
Responsible Party: Sponsor
Other Study IDs: LRC 01.002
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Non Metastatic HER2 Positive Breast Cancer
Keywords: HER2 positive; Breast cancer; non metastatic; Neoadjuvant therapy; Algerian women; Subcutaneous trastuzumab-pertuzumab; pathologic complete response
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to find out how effective and well-tolerated the subcutaneous form of trastuzumab-pertuzumab (known as Phesgo) is when given before surgery (neoadjuvant treatment) to Algerian women with early stage, HER2-positive breast cancer.

The study will take place in three oncology centers in Algeria (Blida, Aïn Defla, Médéa) and include around 70 adult women diagnosed with non-metastatic HER2-positive breast cancer. Participants will receive Phesgo along with standard chemotherapy over about 18 weeks, followed by surgery.

The main goal is to measure how many women achieve complete destruction of invasive cancer in the breast and nearby lymph nodes (pathological complete response, pCR). We will also look at other outcomes such as how many women can keep their breast, any side effects, quality of life, satisfaction with treatment, and factors that might predict response.

Results from this real-world study will help assess whether Phesgo can simplify treatment delivery, reduce hospital burden, and improve care access in Algeria where healthcare resources are often stretched.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 19 years or older.
* Histologically confirmed HER2-positive breast cancer (by immunohistochemistry and/or in situ hybridization), non-metastatic.
* Candidate for neoadjuvant therapy according to local clinical practice.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Left ventricular ejection fraction (LVEF) ≥ 50%.
* Signed written informed consent.

Exclusion Criteria:

* Evidence of distant metastases.
* Prior anti-HER2 therapy.
* Known contraindications to trastuzumab or pertuzumab.
* Pregnancy or breastfeeding.
* Disease progression during neoadjuvant treatment (if already started).
* Refusal of surgery.
* Withdrawal of consent.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients diagnosed with HER2-positive, non-metastatic breast cancer and eligible for neoadjuvant therapy according to local clinical practice in Algeria. Participants will be recruited from three oncology centers: Anti Cancer Center of Blida, public hospital of Aïn Defla, and public hospital of Médéa.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | At the time of surgery, approximately 18-24 weeks after the start of neoadjuvant treatment.
  The proportion of participants with no residual invasive cancer in the breast and axillary lymph nodes after completion of neoadjuvant therapy, defined as ypT0/Tis ypN0 according to standard pathological assessment.
  Pathological evaluation will be performed on surgical specimens by certified pathologists following local and international guidelines.

SECONDARY OUTCOMES:
Breast-Conserving Surgery Rate | At the time of surgery, approximately 18-24 weeks after the start of neoadjuvant treatment.
  Proportion of participants undergoing breast-conserving surgery after completion of neoadjuvant therapy. Determined from surgical records.
Incidence of Adverse Events | From first dose of study treatment until 30 days after last dose (approximately 20-22 weeks).
  Frequency and severity of treatment-related adverse events, graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version in use at study initiation.
Patient Satisfaction With Treatment | Post-surgery (approximately 24-28 weeks after treatment initiation).
  Proportion of participants reporting satisfaction with subcutaneous administration of trastuzumab-pertuzumab (Phesgo), as assessed by a study-specific satisfaction questionnaire.
Predictive Factors of Response | From baseline to surgery (approximately 18-24 weeks after treatment initiation).
  Association between clinical, pathological, and biological characteristics (including biomarkers) and pathological complete response.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical oncology department - Anti Cancer Center of Blida, Blida, Algeria